CLINICAL TRIAL: NCT05418946
Title: Observational Retrospective Cohort Study to Evaluate the Benefits, Documented in Experimental Settings, of Treatment With DAPAGLIFLOZIN in Normal Clinical Practice, in Subjects With Type 2 Diabetes
Brief Title: The Effects of Dapagliflozin in Normal Clinical Practice in T2D
Acronym: PRECARE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Paolo Fiorina, MD, Professor, University of Milan
Other Study IDs: 2022002
Record Dates: First submitted 2022-04-13; First posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Type 2 Diabetes
Keywords: Dapagliflozin; Renal function
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Treatment group: Patient in treatment with Dapagliflozin 10 mg/day
  Interventions: Drug: Dapagliflozin 10mg

INTERVENTIONS:
Drug: Dapagliflozin 10mg — Treatment of T2D and cardio-renal prevention
  Other Names: Forxiga

SUMMARY:
The aim of the study is to evaluate the benefits, documented in experimental settings, of treatment with Dapagliflozin in subjects with type 2 diabetes in normal clinical practice.

The type of study does not involve immediate risks or direct benefits for the subjects taking part in it. The potential benefits for clinicians and healthcare systems are: greater knowledge of diabetic disease and the study of new treatment options. However, the analysis of the data will allow us to better identify which patients benefit most from treatment with Dapagliflozin.

DETAILED DESCRIPTION:
An observational, multicentric, non-interventional, non-profit, single-arm, retrospective prospective study is proposed, aimed at investigating the therapeutic efficacy at 4 months of a treatment with Dapagliflozin® in subjects with type 2 diabetes mellitus belonging to the Lombard centers who joined the study.

Patient recruitment will be carried out at the Unit of Endocrine Diseases and Diabetology in the L. Sacco, Fatebenefratelli and Oftalmico e Macedonio Melloni hospitals, directed by Prof. Paolo Fiorina. Upon enrollment, the informed consent signed and dated by the doctor who informed the patient and by the patient himself will be collected as well as the patient's medical and anamnestic data. This study does not foresee that additional diagnostic or monitoring procedures will be implemented on patients outside of normal clinical practice. The duration of the study per patient after enrollment is 6 months.

This study involves the collection of retrospective data (review of patient medical records). The collection of retrospective data will be done to study the clinical characteristics of the patients at the time they started Dapagliflozin®. The study aims to compare the results reported in the literature with the efficacy outcomes in real-life; to this end, the main clinical and biometric parameters of adult patients with type 2 diabetes belonging to the centers that have joined the study and have been on therapy with Dapagliflozin® for at least 4 months will be collected.

By compiling an online database, the parameters and the respective 4-month variations will be entered anonymously and processed in an aggregate manner in compliance with current regulations and regulatory activities for the conduct of observational retrospective studies.

The insertion of the observations will end after 6 months from the authorization.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type II diabetes mellitus, according to ADA indications for at least 3 months
* Males or females> 18 years old
* Stable therapy for at least 3 months with oral hypoglycemic agents / insulin
* Prescription of Dapagliflozin®, according to normal clinical practice and local indications for the prescription / reimbursement of the drug.

Exclusion Criteria:

* Mental incapacity, unavailability or language barriers that preclude adequate understanding or cooperation;
* Diagnosis of type 1 diabetes mellitus, maturity-onset diabetes of the young (MODY), latent autoimmune diabetes in adults (LADA), gestational diabetes mellitus, secondary diabetes mellitus or any other hyperglycemic state other than type 2 diabetes (T2D);
* Women who are pregnant or breastfeeding, or women planning to become pregnant;
* Previous participation in the study. Participation is defined by having given informed consent to the study;
* Participation in another clinical study on T2D that includes any clinical intervention or administration of an investigational drug within 3 months prior to enrollment in the study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: T2D patients who undergone treatment with Dapagliflozin
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Variation in glycated hemoglobin (HbA1c) values (% -point) from baseline to 4 months from enrollment | From baseline to 4 months

SECONDARY OUTCOMES:
Assessment of the change in fasting glycemic control (mg/dl) | From baseline to 4 months
Evaluation of Body Mass Index (BMI) (kg/m2) | From baseline to 4 months
Evaluation of hip and waist circumferences (cm) | From baseline to 4 months
Evaluation of systolic and diastolic blood pressure (mmHg) | From baseline to 4 months
Evaluation of glomerular filtration rate (GFR) (ml/min/1.73m2) | From baseline to 4 months
Evaluation of albuminuria (mg/g creatinine) | From baseline to 4 months
  Albuminuria will be assessed as albumin to creatinine ratio (ACR) which is obtained from the ratio of urinary protein concentration to creatinine in spot urine

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Fiorina, MD, PhD, Principal Investigator — University of Milan, ASST-FBF-Sacco
Locations (1):
- ASST FBF Sacco, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wilding J, Bailey C, Rigney U, Blak B, Kok M, Emmas C. Dapagliflozin therapy for type 2 diabetes in primary care: Changes in HbA1c, weight and blood pressure over 2 years follow-up. Prim Care Diabetes. 2017 Oct;11(5):437-444. doi: 10.1016/j.pcd.2017.04.004. Epub 2017 Jun 2. PMID 28583425
- [Background] Jongs N, Greene T, Chertow GM, McMurray JJV, Langkilde AM, Correa-Rotter R, Rossing P, Sjostrom CD, Stefansson BV, Toto RD, Wheeler DC, Heerspink HJL; DAPA-CKD Trial Committees and Investigators. Effect of dapagliflozin on urinary albumin excretion in patients with chronic kidney disease with and without type 2 diabetes: a prespecified analysis from the DAPA-CKD trial. Lancet Diabetes Endocrinol. 2021 Nov;9(11):755-766. doi: 10.1016/S2213-8587(21)00243-6. Epub 2021 Oct 4. PMID 34619106
- [Background] Wiviott SD, Raz I, Bonaca MP, Mosenzon O, Kato ET, Cahn A, Silverman MG, Zelniker TA, Kuder JF, Murphy SA, Bhatt DL, Leiter LA, McGuire DK, Wilding JPH, Ruff CT, Gause-Nilsson IAM, Fredriksson M, Johansson PA, Langkilde AM, Sabatine MS; DECLARE-TIMI 58 Investigators. Dapagliflozin and Cardiovascular Outcomes in Type 2 Diabetes. N Engl J Med. 2019 Jan 24;380(4):347-357. doi: 10.1056/NEJMoa1812389. Epub 2018 Nov 10. PMID 30415602
- [Background] Kato ET, Silverman MG, Mosenzon O, Zelniker TA, Cahn A, Furtado RHM, Kuder J, Murphy SA, Bhatt DL, Leiter LA, McGuire DK, Wilding JPH, Bonaca MP, Ruff CT, Desai AS, Goto S, Johansson PA, Gause-Nilsson I, Johanson P, Langkilde AM, Raz I, Sabatine MS, Wiviott SD. Effect of Dapagliflozin on Heart Failure and Mortality in Type 2 Diabetes Mellitus. Circulation. 2019 May 28;139(22):2528-2536. doi: 10.1161/CIRCULATIONAHA.119.040130. Epub 2019 Mar 18. PMID 30882238